CLINICAL TRIAL: NCT05196334
Title: Pharmacotyping of Patient-derived Pancreatic Cancer Organoids From Endoscopic Ultrasound-guided Biopsy as a Tool for Predicting Oncological Response
Brief Title: Pharmacotyping of Pancreatic Patient-derived Organoids
Status: Recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pia Klausen, Principal Investigator, Herlev Hospital
Other Study IDs: Pancreatic organoid protocol
Record Dates: First submitted 2021-10-14; First posted 2022-01-19 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer
Keywords: organoid; personalized medicine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — organoid cultures will be derived from endoscopic ultrasound-guided fine needle biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
EUS-FNB samples will be used for organoid cultures, which will be co-cultured with cancer associated fibroblasts derived from the surrounding stroma of the lesion. The organoid cultures will be used for pharmacotyping using relevant chemotherapeutic agents used in the clinic, and the organoid's response compared with the patient's response.

DETAILED DESCRIPTION:
Aim: To use organoids cultured from diagnostic endoscopic ultrasound (EUS)-guided fine needle biopsy (FNB) samples from patients with pancreatic ductal adenocarcinoma (PDAC) for pharmacotyping.

Patients will be included at Herlev Hospital. EUS-FNB will be performed using a standard 19 or 22-gauge FNB needle. Oncological treatment administration and evaluation of treatment response will be performed by physicians at the Department of Oncology, Herlev Hospital as per current standard of care. Following EUS-FNB procedure, the tissue is immediately transferred to basal medium and epithelial cells as well as CAFs released by digestion and epithelial cells cultured in Matrigel. Following expansion of the organoids and prior to pharmacotyping, next generation sequencing (NGS) analysis will be performed on both the baseline and the organoid sections to validate if the outgrown organoids correspond to the cancer cells from the baseline sample.

Organoid co-cultures are exposed to six to ten different drug concentrations ranging from 10-12-10-4 M (depending on the individual drug properties). Systemic agents and combinations used in the standard clinical practise will be used. Computed tomography (CT) scan of the thorax and abdomen are performed at baseline (within 28 days prior to first study drug administration) to assess efficacy of the drugs in patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histopathological confirmation of PDAC and planned standard first-line treatment prior to entering this study OR Patients suspected of primary locally advanced, non-metastatic PDAC based on cross-sectional imaging undergoing diagnostic standard of care (SOC) EUS-FNB procedure
* Age > 18 years and older
* Life expectancy greater than 3 months
* ECOG/WHO Performance Status (PS) 0-1
* Patients must have normal organ and marrow function as defined below:
* White blood cell count (WBC) ≥ 3 x 10⁹/L
* Platelet count ≥ 100 x 10⁹/L
* Serum bilirubin ≤1.5 x upper limit of normal (ULN) (patients with Gilbert's Syndrome must have a total bilirubin ≤ 50 mmol/L)
* PP ≥ 40 or INR ≤ 1.5
* Serum creatinine ≤ 1.5 x ULN or CrCl ≥ 40 mL/min (using the Cockcroft-Gault formula)

Exclusion Criteria:

* Contraindications for nurse administered propofol sedation (NAPS)
* Contraindications for EUS-FNB procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histopathological confirmation of pancreatic ductal adenocarcimona, ineligible for surgery, planned to start standard first line treatment
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of organoid's response to therapy | Organoid co-cultures will be established and pharmacotyped in a timeframe of 2-4 weeks.
  Response of patient derived organoids to standard chemotherapeutic agents used for treatment of patients with pancreatic cancer
Validation of patient's response to therapy | 3 months follow up
  Computed tomography (CT) scan of the thorax and abdomen are performed at baseline (within 28 days prior to first study drug administration) to assess efficacy of the drugs in patients.
Comparison between organoid's and patient's response | 4 months
  The response measured in the pharmacoscreen of organoids will be compared with the patient's response

CONTACTS AND LOCATIONS:
Overall Officials: Pia H Klausen, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Endoscopy Unit, Herlev Hospital, Herlev, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Boj SF, Hwang CI, Baker LA, Chio II, Engle DD, Corbo V, Jager M, Ponz-Sarvise M, Tiriac H, Spector MS, Gracanin A, Oni T, Yu KH, van Boxtel R, Huch M, Rivera KD, Wilson JP, Feigin ME, Ohlund D, Handly-Santana A, Ardito-Abraham CM, Ludwig M, Elyada E, Alagesan B, Biffi G, Yordanov GN, Delcuze B, Creighton B, Wright K, Park Y, Morsink FH, Molenaar IQ, Borel Rinkes IH, Cuppen E, Hao Y, Jin Y, Nijman IJ, Iacobuzio-Donahue C, Leach SD, Pappin DJ, Hammell M, Klimstra DS, Basturk O, Hruban RH, Offerhaus GJ, Vries RG, Clevers H, Tuveson DA. Organoid models of human and mouse ductal pancreatic cancer. Cell. 2015 Jan 15;160(1-2):324-38. doi: 10.1016/j.cell.2014.12.021. Epub 2014 Dec 31. PMID 25557080
- [Background] Tiriac H, Bucobo JC, Tzimas D, Grewel S, Lacomb JF, Rowehl LM, Nagula S, Wu M, Kim J, Sasson A, Vignesh S, Martello L, Munoz-Sagastibelza M, Somma J, Tuveson DA, Li E, Buscaglia JM. Successful creation of pancreatic cancer organoids by means of EUS-guided fine-needle biopsy sampling for personalized cancer treatment. Gastrointest Endosc. 2018 Jun;87(6):1474-1480. doi: 10.1016/j.gie.2017.12.032. Epub 2018 Jan 9. PMID 29325707
- [Background] Seppala TT, Zimmerman JW, Sereni E, Plenker D, Suri R, Rozich N, Blair A, Thomas DL 2nd, Teinor J, Javed A, Patel H, Cameron JL, Burns WR, He J, Tuveson DA, Jaffee EM, Eshleman J, Szabolcs A, Ryan DP, Ting DT, Wolfgang CL, Burkhart RA. Patient-derived Organoid Pharmacotyping is a Clinically Tractable Strategy for Precision Medicine in Pancreatic Cancer. Ann Surg. 2020 Sep 1;272(3):427-435. doi: 10.1097/SLA.0000000000004200. PMID 32657929
- [Background] Tiriac H, Belleau P, Engle DD, Plenker D, Deschenes A, Somerville TDD, Froeling FEM, Burkhart RA, Denroche RE, Jang GH, Miyabayashi K, Young CM, Patel H, Ma M, LaComb JF, Palmaira RLD, Javed AA, Huynh JC, Johnson M, Arora K, Robine N, Shah M, Sanghvi R, Goetz AB, Lowder CY, Martello L, Driehuis E, LeComte N, Askan G, Iacobuzio-Donahue CA, Clevers H, Wood LD, Hruban RH, Thompson E, Aguirre AJ, Wolpin BM, Sasson A, Kim J, Wu M, Bucobo JC, Allen P, Sejpal DV, Nealon W, Sullivan JD, Winter JM, Gimotty PA, Grem JL, DiMaio DJ, Buscaglia JM, Grandgenett PM, Brody JR, Hollingsworth MA, O'Kane GM, Notta F, Kim E, Crawford JM, Devoe C, Ocean A, Wolfgang CL, Yu KH, Li E, Vakoc CR, Hubert B, Fischer SE, Wilson JM, Moffitt R, Knox J, Krasnitz A, Gallinger S, Tuveson DA. Organoid Profiling Identifies Common Responders to Chemotherapy in Pancreatic Cancer. Cancer Discov. 2018 Sep;8(9):1112-1129. doi: 10.1158/2159-8290.CD-18-0349. Epub 2018 May 31. PMID 29853643
- [Background] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484
- [Background] Broutier L, Mastrogiovanni G, Verstegen MM, Francies HE, Gavarro LM, Bradshaw CR, Allen GE, Arnes-Benito R, Sidorova O, Gaspersz MP, Georgakopoulos N, Koo BK, Dietmann S, Davies SE, Praseedom RK, Lieshout R, IJzermans JNM, Wigmore SJ, Saeb-Parsy K, Garnett MJ, van der Laan LJ, Huch M. Human primary liver cancer-derived organoid cultures for disease modeling and drug screening. Nat Med. 2017 Dec;23(12):1424-1435. doi: 10.1038/nm.4438. Epub 2017 Nov 13. PMID 29131160
- [Background] Votanopoulos KI, Mazzocchi A, Sivakumar H, Forsythe S, Aleman J, Levine EA, Skardal A. Appendiceal Cancer Patient-Specific Tumor Organoid Model for Predicting Chemotherapy Efficacy Prior to Initiation of Treatment: A Feasibility Study. Ann Surg Oncol. 2019 Jan;26(1):139-147. doi: 10.1245/s10434-018-7008-2. Epub 2018 Nov 9. PMID 30414038
- [Background] Ohlund D, Handly-Santana A, Biffi G, Elyada E, Almeida AS, Ponz-Sarvise M, Corbo V, Oni TE, Hearn SA, Lee EJ, Chio II, Hwang CI, Tiriac H, Baker LA, Engle DD, Feig C, Kultti A, Egeblad M, Fearon DT, Crawford JM, Clevers H, Park Y, Tuveson DA. Distinct populations of inflammatory fibroblasts and myofibroblasts in pancreatic cancer. J Exp Med. 2017 Mar 6;214(3):579-596. doi: 10.1084/jem.20162024. Epub 2017 Feb 23. PMID 28232471
- [Background] Seino T, Kawasaki S, Shimokawa M, Tamagawa H, Toshimitsu K, Fujii M, Ohta Y, Matano M, Nanki K, Kawasaki K, Takahashi S, Sugimoto S, Iwasaki E, Takagi J, Itoi T, Kitago M, Kitagawa Y, Kanai T, Sato T. Human Pancreatic Tumor Organoids Reveal Loss of Stem Cell Niche Factor Dependence during Disease Progression. Cell Stem Cell. 2018 Mar 1;22(3):454-467.e6. doi: 10.1016/j.stem.2017.12.009. Epub 2018 Jan 11. PMID 29337182
- [Result] Engholm G, Ferlay J, Christensen N, Bray F, Gjerstorff ML, Klint A, Kotlum JE, Olafsdottir E, Pukkala E, Storm HH. NORDCAN--a Nordic tool for cancer information, planning, quality control and research. Acta Oncol. 2010 Jun;49(5):725-36. doi: 10.3109/02841861003782017. PMID 20491528